CLINICAL TRIAL: NCT05489445
Title: Evaluating KODEX-EPD Electrophysiology Mapping During Cryoballoon Pulmonary Vein Isolation
Brief Title: All Inclusive Kodex - EPD Study
Status: Terminated | Type: Observational
Why Stopped: Sponsor closed the product line.
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Wilber Su, Clinical Associate Professor, Cardiology, University of Arizona
Other Study IDs: 2103636199
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation
Keywords: irregular heart beat; rapid heart beat; Cryoballoon ablation; Cardiac Imaging; 3D mapping; Afib ablation; Atrial fibrillation; Pulmonary vein isolation; 3D mapping of the heart
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Tachycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing EP: Patients already clinically indicated for undergoing catheter-based eletrophysiological intervention, in which the FDA approved medical device KODEX-EPD system will be used.
  Interventions: Device: KODEX - EPD

INTERVENTIONS:
Device: KODEX - EPD — A patient that is already clinically indicated to undergo cryoballoon ablation for atrial fibillation will use the The KODEX - EPD™ Cardiac Imaging and Navigation electrophysiological (EP) System. This is an imaging system which allows the physician real-time visualization of the catheters in a patients heart during the procedure, as well as display of cardiac images of the patients heart in a number of different formats. The KODEX - EPD system used in this study is cleared for commercial use by the FDA and therefore, it's use in this study constitutes as standard clinical use.

SUMMARY:
This is a post-market, prospective, observational study to evaluate the accuracy of KODEX 3D-imaging. The research study will collect pre-operative and post-operative cardiac imaging data from adult arrhythmia patients who are already undergoing catheter-based electrophysiological (EP) intervention (ablation procedures) using the FDA approved medical device KODEX - EPD™ system.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is among the most prevalent arrhythmias in the world affecting approximately 1.5-2.0% of the general population. The age of patients with AF is steadily rising and now averages between 75 and 85 years of age. AF is associated with a five-fold risk of stroke, a three-fold incidence of congestive heart failure, and higher mortality.

Symptoms arise from the rapid, irregular rhythm as well as the loss of cardiac pump function related to uncoordinated atrial contractions. These uncoordinated contractions also allow blood to pool in the atria and may ultimately lead to thromboembolism and stroke. AF is characterized by a chaotic contraction of the atrium in which an electrocardiogram (ECG) recording is necessary to diagnose the arrhythmia . The diagnosis requires an ECG demonstrating: (1) Irregular RR intervals (in the absence of complete AV block), (2) no distinct P waves on the surface ECG, and (3) an atrial cycle length (when visible) that is usually variable and less than 200 milliseconds.

Initial therapy of atrial fibrillation is usually directed toward reversion to and maintenance of sinus rhythm through drug therapy. However, drug therapy can be associated with a number of unwanted effects such as proarrhythmia, long-term ineffectiveness, and even an increase in mortality, especially in those with impaired ventricular function. In the treatment of Atrial Fibrillation (AF) catheter ablation is considered superior regarding freedom of arrhythmia recurrence compared to anti-arrhythmic drug therapy. , , . Intracardiac ablation has been developed using a technique of pulmonary vein isolation (PVI) to disconnect the rapid firing of the pulmonary veins from the rest of the left atrium. Current guidelines recommend PVI by means of catheter ablation as treatment for symptomatic drug-refractory paroxysmal AF . Radiofrequency and cryoballoon catheters are the most frequently utilized ablation modalities. It has been demonstrated that cryoballoon ablation is non-inferior to radiofrequency ablation with respect to efficacy for the treatment of patients with drug-refractory paroxysmal AF, and there were no differences with regard to overall safety.

Current catheter-based therapy utilizes cardiac 3D mapping and navigation systems that were introduced more than 20 years ago and allow location of the ablation device within a reconstruction of the heart anatomy , , , . However, technical limitations specific to each available 3D mapping system, such as variability in catheter tip location sensing, alternating location reliability throughout the procedure, and the use of costly specialized catheters and additional hardware (e.g. magnets placed under the operating table, pose limitations of these systems. Furthermore, all available systems provide only an estimate of each individual anatomy, as they do not provide high-quality, real-time visualization of anatomical structures, but merely a low-resolution reconstruction. In order to obtain more information and a precisely detailed anatomy, time consuming and often costly additional imaging such as fluoroscopy, angiography, echocardiography and even pre-procedural computer tomography (CT) and magnetic resonance imaging (MRI) is required in many cases.

In conclusion the current procedures are relatively long, considered highly complex and require substantial expertise. In addition, specialized catheters and additional hardware are required. The manufacturer has identified these challenges and has developed the KODEX - EPD system to address them.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Documented atrial fibrillation

Exclusion Criteria:

* Prior history left atrial catheter ablation and/or surgical maze procedure
* Pregnancy as confirmed with positive blood test at index procedure
* Prior history of congenital heart condition resulting in anomalous pulmonary vein anatomy
* left ventricular ejection fraction less than or equal to 35%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will be selected from patients undergoing EP study at BUMCP in either an inpatient or outpatient setting, then followed in the Banner Heart Institute.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Acute PVI during index procedure. | During EP
  Use of segmental approach versus "one-shot" balloon application.
Long term efficacy | Up to 3 years post index procedure
  Efficacy of PVI post index PVI

SECONDARY OUTCOMES:
Exploratory | Up to 5 years after first enrolled subject
  Use of KODEX-EPD tissue characteristics to predict need for the segmental approach with cryoballoon

CONTACTS AND LOCATIONS:
Locations (1):
- Banner - University Medical Center, Phoenix campus, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers.

REFERENCES:
- [Background] Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, Hindricks G, Kirchhof P; ESC Committee for Practice Guidelines-CPG; Document Reviewers. 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation--developed with the special contribution of the European Heart Rhythm Association. Europace. 2012 Oct;14(10):1385-413. doi: 10.1093/europace/eus305. Epub 2012 Aug 24. No abstract available. PMID 22923145
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2017 Oct;14(10):e275-e444. doi: 10.1016/j.hrthm.2017.05.012. Epub 2017 May 12. No abstract available. PMID 28506916
- [Background] European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery; Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Eur Heart J. 2010 Oct;31(19):2369-429. doi: 10.1093/eurheartj/ehq278. Epub 2010 Aug 29. No abstract available. PMID 20802247
- [Background] Calkins H, Reynolds MR, Spector P, Sondhi M, Xu Y, Martin A, Williams CJ, Sledge I. Treatment of atrial fibrillation with antiarrhythmic drugs or radiofrequency ablation: two systematic literature reviews and meta-analyses. Circ Arrhythm Electrophysiol. 2009 Aug;2(4):349-61. doi: 10.1161/CIRCEP.108.824789. Epub 2009 Jun 2. PMID 19808490
- [Background] Wilber DJ, Pappone C, Neuzil P, De Paola A, Marchlinski F, Natale A, Macle L, Daoud EG, Calkins H, Hall B, Reddy V, Augello G, Reynolds MR, Vinekar C, Liu CY, Berry SM, Berry DA; ThermoCool AF Trial Investigators. Comparison of antiarrhythmic drug therapy and radiofrequency catheter ablation in patients with paroxysmal atrial fibrillation: a randomized controlled trial. JAMA. 2010 Jan 27;303(4):333-40. doi: 10.1001/jama.2009.2029. PMID 20103757
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Kuck KH, Ernst S, Cappato R, Braun E, Lang M, Ben-Haim SA, Hebe J, Ouyang F, Khanedani A, Antz M, Volkmer M. Nonfluoroscopic endocardial catheter mapping of atrial fibrillation. J Cardiovasc Electrophysiol. 1998 Aug;9(8 Suppl):S57-62. PMID 9727677
- [Background] Ben-Haim SA, Osadchy D, Schuster I, Gepstein L, Hayam G, Josephson ME. Nonfluoroscopic, in vivo navigation and mapping technology. Nat Med. 1996 Dec;2(12):1393-5. doi: 10.1038/nm1296-1393. No abstract available. PMID 8946843
- [Background] Stevenson WG, Delacretaz E, Friedman PL, Ellison KE. Identification and ablation of macroreentrant ventricular tachycardia with the CARTO electroanatomical mapping system. Pacing Clin Electrophysiol. 1998 Jul;21(7):1448-56. doi: 10.1111/j.1540-8159.1998.tb00217.x. PMID 9670190
- [Background] Gepstein L, Hayam G, Ben-Haim SA. A novel method for nonfluoroscopic catheter-based electroanatomical mapping of the heart. In vitro and in vivo accuracy results. Circulation. 1997 Mar 18;95(6):1611-22. doi: 10.1161/01.cir.95.6.1611. PMID 9118532
- [Background] Maurer T, Mathew S, Schluter M, Lemes C, Riedl J, Inaba O, Hashiguchi N, Reissmann B, Fink T, Rottner L, Rillig A, Metzner A, Ouyang F, Kuck KH. High-Resolution Imaging of LA Anatomy Using a Novel Wide-Band Dielectric Mapping System: First Clinical Experience. JACC Clin Electrophysiol. 2019 Nov;5(11):1344-1354. doi: 10.1016/j.jacep.2019.06.020. Epub 2019 Aug 28. PMID 31753443